CLINICAL TRIAL: NCT06033924
Title: Telehealth Delivered Home-based Walking for Vets With Peripheral Artery Disease (TREK-PAD)
Brief Title: Telehealth Delivered Home-based Walking for Vets With Peripheral Artery Disease
Acronym: TREK-PAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E3965-R
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral artery disease; physical activity; quality of life
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Internet-based Walking Program (Experimental): Internet pages allow participants to see step-count goals, progress over time and access to walking tips
  Interventions: Behavioral: Walking Program: Internet-based
- Telehealth Counseling Walking Program (Experimental): Telehealth sessions allow participants review step-count goals, progress over time and access to walking tips with the study coordinator
  Interventions: Behavioral: Walking Program: Telehealth-based

INTERVENTIONS:
Behavioral: Walking Program: Internet-based — Internet pages allow participants to see step-count goals, progress over time and access to walking tips for 12 weeks. Among participants who do not increase their step counts (>15%), these non-responders will be rerandomized to received the combination of internet and telehealth or either along for an additional 12-weeks (total intervention time is 24-weeks). A follow-up phase of 12-weeks will be completed for a total participant duration of 36 weeks.
  Arms: Internet-based Walking Program
Behavioral: Walking Program: Telehealth-based — Telehealth sessions allow participants review step-count goals, progress over time and access to walking tips with the study coordinator for 12 weeks. Among participants who do not increase their step counts (>15%), these non-responders will be rerandomized to received the combination of internet and telehealth or either along for an additional 12-weeks (total intervention time is 24-weeks). A follow-up phase of 12-weeks will be completed for a total participant duration of 36 weeks.
  Arms: Telehealth Counseling Walking Program

SUMMARY:
Walking is beneficial for adults with peripheral arterial disease. Benefits include the ability to walk for longer periods and general well being (quality of life). This study will look at two types of delivery methods for a home-based walking program. The walking program includes step count goals, information on healthy walking and motivational messages. The two delivery methods include a web-based delivery and an telehealth delivery. Participants are randomized to either one of the delivery methods or usual care. After 12 weeks participants in the web based or telehealth based groups maybe re-randomized to receive a combination of both web-based and telehealth for a second 12 week period. After 24 weeks, everyone is followed for an additional 12 weeks, so the total time a participant is in the study is 36 weeks. At baseline, 12, 24 and 36 weeks the investigators ask participant to walk (slowly) on a treadmill, perform a six-minute walk test, and several questionnaires on quality of life. Vouchers are provided at each study visit. All participants who complete the study also keep their pedometer.

DETAILED DESCRIPTION:
The objective of this study is to evaluate two delivery methods of home-based walking among Veterans with PAD. The investigators will use an innovative sequential multiple assignment, randomized trial (SMART) design to compare a web-based delivered (WBD) walking program and a video telehealth delivered (VTD) walking program versus usual care among 225 Veterans with peripheral arterial disease (PAD) in three sites (Birmingham AL, Palo Alto CA, and Aurora CO).

This trial has two study aims and one exploratory aim. Aim 1 is to evaluate the efficacy of two remote delivery methods to increase maximal walking distance, pain-free walking distance, and health-related quality of life (HRQOL) compared to baseline, among Veterans with PAD. The investigators hypothesize that at 12-weeks, participants initially randomized to the WBD program and the VTD program will have greater improvement in maximal walking distance (primary outcome) compared to usual care (UC). Furthermore, this improvement (for both WBD and VTD) will be sustained at 24-weeks compared to UC, and at 12- and 24-weeks, both the WBD program and the VTD program will produce greater improvement in pain-free walking distance and HRQOL compared to UC.

Study aim 2 is to evaluate the efficacy of the combination of WBD with a VTD walking program among Veterans who do not respond to their initial assignment. The investigators hypothesize that at 24- and 36-weeks, the combination of WBD+VTD will produce greater improvements in maximal walking distance (from second randomization at 12-weeks) compared to either WBD or VTD alone.

The exploratory aim is to compare the efficacy of WBD and VTD and to examine factors associated (age, race/ethnicity, rural residency, engagement, co-morbidities (including CVD risk), and PAD symptoms/severity) with initial response to WBD and VTD to identify the most effective strategy to increase mobility in Veterans with PAD.

Design & Outcomes: Using a randomized control trial design with sequential multiple assignments, participants will be randomized to 1 of 3 arms; a web-based delivered (WBD) walking program, (ii) a video telehealth delivered (VTD) walking program, or (iii) usual care (UC) only.

Intervention & Duration: The interventions include i) the web-based delivered (WBD) walking program and (ii) the video telehealth delivered (VTD) walking program. All participants, irrespective of study assignment, will receive two in-person visits with an exercise physiologist prior to randomization. After 12 weeks, participants in the WBD arm who do not respond will be further randomized to receive WBD + VTD or WBD only, and participants in the VTD arm who do not respond will be further randomized to receive VTD + WBD or VTD only. Nonresponse will be defined as a <15% increase in maximal walk distance compared to baseline (measured with a validated treadmill protocol at 12 weeks). The interventions will then continue for an additional 12 weeks (for a total of 24 weeks of the intervention). After the 24-week visit, participants will be followed for an additional 12 weeks to examine longer-term responses for a total participant study duration of 36 weeks. A third arm will include participants randomized to usual care (UC)

Outcomes include maximal and pain-free walking distance, and health-related quality of life (HRQOL) will be measured at all visits (i.e., baseline, 12-, 24-, and 36 weeks). The primary outcome of interest is a change in maximal walking distance from baseline to 12 weeks. Secondary outcomes include the change in maximal walking distance at 24 and 36 weeks and a change in pain-free walking distance and HRQOL at 12-, 24- and 36 weeks. Primary and secondary outcomes will be measured in all participants.

Sample Size & Population: A total of 225 Veterans with PAD will be enrolled. Men and women Veterans with atherosclerosis of arteries/arterial bed(s) of the lower extremities (including aortoiliac, aortofemoral, iliac, femoral, femoropopliteal, and popliteal), who report claudication symptoms, will be potentially eligible for this study. Diagnosis of lower extremity PAD due to atherosclerosis is defined as an ankle-brachial index (ABI) < 0.9 in at least one lower extremity or evidence of critical stenosis (> 70%) in at least one vascular territory below the waist by CT angiography, MRI, or peripheral angiogram. Patients with PAD due to non-atherosclerotic etiologies, such as trauma, entrapment syndromes, or congenital abnormalities, are excluded. Vulnerable populations, including children, pregnant women, fetuses, neonates, abortuses, anyone with impaired decision-making capacity, cancer subjects, students, employees, prisoners, or international participants will not be enrolled. Only adults with PAD will be eligible; therefore, the investigators will exclude healthy volunteers. PAD is diagnosed during adulthood; therefore, children are unlikely to have the condition. The investigators will not limit enrollment by sex or race/ethnicity. Potential participants will be recruited through cardiology and vascular clinics. After the eligibility screening is complete and all participant questions have been answered, the participant will provide written informed consent prior to study enrollment.

Data collection: Data will be collected at four study visits. Baseline Visit (Visit 1): All potential subjects will be screened to confirm initial eligibility, including a review of the EMR to confirm a diagnosis of PAD and absence of exclusion criteria. At the baseline visit, all questions from the potential participant will be answered, and final confirmation of eligibility will be completed. Thereafter, written informed consent will be obtained. Data to be collected at this visit include baseline demographics, medical history, measures of physical function (maximal and pain-free walking distance and six-minute walk distance [6MWD]), and survey data (e.g., HRQOL). PAD symptoms are collected through pain-free walking distance, the PAQ survey, and Rutherford classification for claudication. The primary outcome of maximal walking distance will be measured using a validated protocol.

Participants, regardless of study arm (including the controls), will receive 2 coaching sessions with an exercise physiologist to review the walking protocol. The coaching will be based on guidelines recommendations for walking programming among adults with claudication associated with PAD. This includes advice to walk until claudication symptoms occur at which time the participant briefly rests until symptoms resolve; if pain-free, the participants can continue walking at a comfortable pace. This will be repeated for the 40 to 50 minutes of exercise, although participants may not be able to walk for 30 minutes at the start of the program, they will be encouraged to build to this duration. Participants will be asked to perform at least three sessions per week for a total of 48 sessions over 16-weeks. This method of walking till claudication occurs is an important component of PAD interventions, with evidence to support greater improvements in maximal walking distance with higher intensity walking behaviors.

Randomization: Randomization will occur at the baseline visit, after eligibility is confirmed and consent is obtained. Permuted block randomization, with a block-sizes of 3 and 6, will be used, and a computer-generated randomization list will be used to assign participants to one of the three study arms. The randomization will not be stratified by clinical, demographic, or socioeconomic factors; these factors will be accounted for in the statistical analysis. Although the investigators are unable to blind participants to treatment arm, personnel completing all study assessments will remain blinded to randomized assignment.

Blinding: As with most behavioral interventions, participants cannot be blinded to treatment assignment. However, all assessments will be conducted by study staff blinded to treatment assignment. The PIs will also be blinded to participant assignment as well. Participants will be reminded not to discuss which intervention they are randomized to prior to each study visit.

Study Visits 2-4: All study participants (including controls) will return for study visits at 12-, 24- and 36-weeks. Participants will complete the same assessments performed at Visit 1. Any changes to medical history, including healthcare utilization (e.g., hospitalization), will be reviewed at each visit. Measures of physical function will be collected (maximal and pain-free walking distance), and surveys to measure HRQOL, PAD symptoms, and non-walking physical activity (i.e., Godin Leisure Time Physical Activity Survey) will be completed by all participants. The participants will be asked about doctor visits or hospitalizations since the prior study visit (in addition to a medical record review). If participants report a hospital admission to an external healthcare system, with the participant's consent, the investigators will request the related medical record for that admission. Changes in medications will also be collected. If a serious event has occurred, the subject will not be cleared for continued participation until the record is reviewed and medical clearance is obtained from their healthcare provider.

Throughout the follow-up, the investigators will collect data on engagement to account for differences in the dosing of the interventions between participants. Participants randomized to the telehealth visits are scheduled to receive, weekly video calls which included tailored messages and weekly tailored step-count goals Participants randomized to the web-based walking program, also receive weekly tailored messages, and weekly tailored step-count goals, through their webpage (with an email reminder). Thus, the dose is similar for each arm. At 12-weeks, non-responders (defined as a <15% increase in maximal walk distance) will be rerandomized to continue with their initial assignment or receive a combination of telehealth calls with the web-based program. The dose of both the telehealth video calls and the web-based program will be unchanged (i.e., weekly). Importantly, the investigators will collect data on engagement, in other words, the number of missed calls for the telehealth component and the frequency of log ins to the web-based platform, to account for potential differences in dosing of the interventions.

During Visit 4, a brief exit interview will be completed by participants. Participants randomized to WBD, VTD, or the combination will be asked about overall satisfaction with the intervention(s), including acceptability, ease of use, method of delivery, and content. The investigators will also ask all participants about facilitators and barriers and solicit suggestions for future programs.

Sources of Data

Maximal & Pain-Free Walking Distance:

Gardener Treadmill Test: Treadmill testing is a Class I recommendation for the assessment of functional limitations and response to therapy. Change in maximal walking distance is the primary outcome, which is measured using the validated protocol developed by Gardener and colleagues. A standard protocol with a constant speed of 2 mph starting at 0% slope and increasing 2% in slope every 2 minutes will be used. This protocol has been well validated and will allow for the assessment of maximal walking distance. Each subject will be instructed to continue to walk until he/she can no longer do so; this distance will be defined as the maximal walking distance (primary outcome). Subjects with claudication symptoms will be instructed to report when they first have symptoms, and this will be recorded as pain-free walking distance. All treadmill testing will be performed by trained exercise physiologists, with a supervising cardiologist, using this standardized method. Blood pressure and heart rate (i.e., ECG) will be monitored prior to and during testing.

Six Minute Walk Distance (6MWD) test has been used to measure physical function in numerous conditions, including PAD. The investigators will use the American Thoracic Society protocol to collect 6MWD in all participants. Given that some prior studies have used the 6MWD, the investigators have opted to collect both measures of maximal walk distance (i.e., treadmill and 6MWD)

Health-related Quality of Life (HRQOL):

The Patient-Reported Outcomes Measurement Information System (PROMIS) is an NIH Common Fund initiative focused on the dynamic assessment of patient-reported outcome measures of HRQOL. PROMIS includes item banks that measure key health symptoms/concepts for both the general population and several chronic conditions. These item banks include assessment for physical (physical function, fatigue, sleep disturbance, sleep-related impairment, pain behavior, pain intensity, pain interference, and sexual function), emotional (depression, anxiety, anger, self-efficacy, and cognitive function), and social health (ability to participate, satisfaction with social roles and activities, companionship, emotional support, instrumental support, informational support, and social isolation). The investigators propose using the PROMIS-29 profile that includes four questions from each of the seven domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities). The estimated time for completion of the PROMIS-29 is < 4 minutes. In addition, the investigators will use the Short Form 4-item general self-efficacy items that can be completed in < 1 minute. The PROMIS-29 yields scores for each of the domains above and a total score. All scores are on a t distribution (mean 50, standard deviation [SD] 10), with higher scores indicating more of the domain that is being measured. Responsiveness-to-change data for PROMIS have been examined in many chronic conditions, with generally small to moderate 3-month effect sizes (0.23 to 0.83) and moderate to large 12-month effect sizes (0.63 to 1.14; effect sizes were calculated as mean change divided by SD at baseline).

Participants will also complete the Peripheral Artery Questionnaire (PAQ), a disease-specific HRQOL measure that is reliable in patients with PAD and has excellent construct validity. The PAQ has seven domains and 20 items that are internally reliable (Cronbach = 0.80 to 0.94) and have acceptable test-retest reliability. Domains include physical limitation, symptoms, symptom stability, social limitation, treatment satisfaction, and a summary score. The average time for completion is < 4 minutes. When used before and after the intervention, such as revascularization, the instrument is sensitive to change and is more sensitive to clinical change than either the SF 36 or the Walking Impairment Questionnaire.

Demographics, Clinical Factors & Cardiovascular Risk Factors Demographic and clinical characteristics: Demographic factors (race/ethnicity, age, and sex), information on medical history (including medications). Comorbidities will include diabetes, hypertension, CVD events (e.g., myocardial infarction, coronary revascularization, heart failure hospitalization and stroke), CKD, lung disease, and smoking history). Social determinants of health characteristics (education, income, health literacy). PAD severity (ABI and anatomic location). Physiologic parameters (blood pressure, heart rate, and body mass index). These variables will be collected for use in multivariate models and to identify factors associated with response to the intervention. These will be collected at baseline with updates/changes assessed at follow-up visits, as appropriate.

Self Determination Theory (SDT) Constructs measured with:

Modifiable SDT constructs will be collected for inclusion in multivariate models and will be important factors for understanding the efficacy of the delivery modes (WBD, VTD) included this trial. Two surveys will be administered. The Psychological Need Satisfaction in Exercise (PNSE) scale; an 18-item validated questionnaire of SDT constructs, includes 3 subscales (6 items/scale) that assess the SDT constructs of perceived competence, autonomy, and relatedness, all within the context of exercise behaviors. The PNSE is commonly used in physical activity trials to measure SDT constructs and their potential mediating role in treatment. The second survey is the Internalized self-regulation or autonomous motivation will be measured with the Treatment Self-Regulation Questionnaire (TSRQ), which includes 6 items asking about respondents' autonomous reasons for engaging in a behavior (i.e., exercise). This instrument has been used widely and demonstrates excellent validity and reliability when applied to a variety of health behaviors and conditions, including physical activity.

Physical Activity The Godin-Shepherd Leisure-Time Physical Activity Questionnaire (GSLTPAQ) will be used to assess non-walking physical activity. The survey assesses the frequency per week of activities from which METS can be calculated. This validated questionnaire is reliable for minority populations.

Step Counts Pedometers: Participants randomized to WBD and VTD study arms can use the pedometers as a motivational tool. However, the investigators will also collect these data to compare with the measure of physical activity noted above. These data will allow us to examine the use of commercially available pedometers for further trials.

Engagement For each intervention and study visit, data on engagement. These data will include number of missed telehealth calls, frequency, and duration of logins to the web platform. For all participants (including controls) any missed study visits and the reasons for absence will be recorded. Lastly, exit interview will be completed by participants, to collect qualitative data on overall satisfaction with the intervention(s), including acceptability, ease of use, method of delivery, and content. The investigators will also ask all participants about facilitators and barriers and solicit suggestions for future programs.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Diagnosis of lower extremity PAD due to atherosclerosis
* Claudication with walking defined as stage 1-3 on the Rutherford Scale
* Medical clearance from the patient's primary care provider or vascular care provider
* Ability to walk at least one city block
* Self-reported sedentary behaviors defined as < 150 minutes per week of physical activity
* Access to a phone and/or email & Internet
* Competent to provide informed consent

Exclusion Criteria:

* Life expectancy of less than six months
* Comorbidities that limit walking to a severe degree (i.e., wheelchair-bound)
* Resident of a nursing home
* Recent enrollment in an exercise program or performing 150 minutes per week or more of exercise
* Planned revascularization or amputation in the next two months
* Recent CVD events (< 3 months) including stroke/TIA, MI, UA, PCI/CABG
* Unstable cardiac conditions (severe valve disease, NYHA class III-IV heart failure, untreated complex congenital heart disease, or complex arrhythmias)
* Current substance abuse
* Psychiatric disorder which limits the patient's ability to follow the study protocol
* Pregnancy
* Inability to speak and read English

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-10-29 (Estimated); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
Change in maximal walking distance | baseline to 12 weeks
  measured using the Gardener-Sinner protocol treadmill test, a validated protocol for measuring maximal and claudication free walking distance among patients with PAD, used in clinical care

SECONDARY OUTCOMES:
Change in maximal walking distance | baseline to 24 weeks
  measured using the Gardener-Sinner protocol treadmill test, a validated protocol for measuring maximal and claudication free walking distance among patients with PAD, used in clinical care
Change in maximal walking distance | baseline to 36 weeks
  measured using the Gardener-Sinner protocol treadmill test, a validated protocol for measuring maximal and claudication free walking distance among patients with PAD, used in clinical care
Change in claudication free walking distance | baseline to 12 weeks
  measured using the Gardener-Sinner protocol treadmill test, a validated protocol for measuring maximal and claudication free walking distance among patients with PAD, used in clinical care
Change in claudication free walking distance | baseline to 24 weeks
  measured using the Gardener-Sinner protocol treadmill test, a validated protocol for measuring maximal and claudication free walking distance among patients with PAD, used in clinical care
Change in claudication free walking distance | baseline to 36 weeks
  measured using the Gardener-Sinner protocol treadmill test, a validated protocol for measuring maximal and claudication free walking distance among patients with PAD, used in clinical care
Change in PAD-specific health-related quality of life | baseline to 12 weeks
  measured using a disease specific validated questionnaire - the Peripheral Artery Questionnaire (PAQ) which uses scale scores of 0 to 100, with high numbers indicating better outcomes.
Change in PAD-specific health-related quality of life | baseline to 24 weeks
  measured using a disease specific validated questionnaire - the Peripheral Artery Questionnaire (PAQ) which uses scale scores of 0 to 100, with high numbers indicating better outcomes.
Change in PAD-specific health-related quality of life | baseline to 36 weeks
  measured using a disease specific validated questionnaire - the Peripheral Artery Questionnaire (PAQ) which uses scale scores of 0 to 100, with high numbers indicating better outcomes.
Change in general health-quality of life | baseline to 12 weeks
  Measuring using the Patient-Reported Outcomes Measurement Information System (PROMIS). The PROMIS 29 include 4 questions form each of 7 domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability's to participate in social roles and activities. The PROMIS-29 yields scores for each of the domains above and a total score. Higher scores represent higher symptoms. For exampled a higher score for fatigue represents greater fatique. A higher total score represents worse quality of life.
Change in general health-quality of life | baseline to 24 weeks
  Measuring using the Patient-Reported Outcomes Measurement Information System (PROMIS). The PROMIS 29 include 4 questions form each of 7 domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability's to participate in social roles and activities. The PROMIS-29 yields scores for each of the domains above and a total score. Higher scores represent higher symptoms. For exampled a higher score for fatigue represents greater fatique. A higher total score represents worse quality of life.
Change in general health-quality of life | baseline to 36 weeks
  Measuring using the Patient-Reported Outcomes Measurement Information System (PROMIS). The PROMIS 29 include 4 questions form each of 7 domains (depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability's to participate in social roles and activities. The PROMIS-29 yields scores for each of the domains above and a total score. Higher scores represent higher symptoms. For exampled a higher score for fatigue represents greater fatique. A higher total score represents worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Jackson, MD, Principal Investigator — Birmingham VA Medical Center, Birmingham, AL
Locations (3):
- United States (3):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No